CLINICAL TRIAL: NCT03283059
Title: Phase III Trial of Octohydroaminoacridine Succinate Tablet for Mild-to-Moderate Alzheimer's Disease: a 26 Weeks, Randomized, Double-blind, Double-dummy, Placebo- and Positive- Parallel Controlled and Extended Single Arm to 54 Weeks Multicentre Study
Brief Title: Octohydroaminoacridine Succinate Tablet for Mild-to-Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Changchun Huayang High-tech Co., Ltd (Industry); Jiangsu Sheneryang High-tech Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHAAS-III
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Octohydroaminoacridine Succinate Tablet (Experimental): Octohydroaminoacridine Succinate Tablet 4mg P.O. tid
  Interventions: Drug: Octohydroaminoacridine Succinate
- Aricept (Active Comparator): Aricept 5mg/day P.O.
  Interventions: Drug: Aricept
- Placebo (Placebo Comparator): Placebo P.O. tid
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Octohydroaminoacridine Succinate — Octohydroaminoacridine Succinate Tablet:4mg P.O. tid
  Arms: Octohydroaminoacridine Succinate Tablet
Drug: Aricept — Aricept 5mg/day, P.O.
  Arms: Aricept
Drug: Placebos — Placebo Tablet: P.O. tid
  Arms: Placebo

SUMMARY:
Inhibition of acetylcholinesterase has been a effective treatment for Alzheimer's disease. Octohydroaminoacridine, a new acetylcholinesterase inhibitor, is a potential treatment for Alzheimer's disease. The investigators conducted a 26 weeks, randomized, double-blind, double-dummy, placebo- and positive- parallel controlled and extended single arm to 54 weeks multicentre phase III clinical trial to investigate the effects of octohydroaminoacridine in patients with mild-to-moderate Alzheimer's disease. Patients were randomized to receive placebo thrice daily, or octohydroaminoacridine 4 mg/TID or ARICEPT 5mg/QD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-85 years (including 50 and 85 years old), male or female;
2. Diagnose probable AD in accordance with the National Institute Aging and Alzheimer's Association (NIA-AA) (2011);
3. Mild-to-moderate AD patients, MMSE 11-26 (including 11 and 26, primary school education subjects from 11 to 22);
4. Hachinski Incheinic Score (HIS) less than 4 points;
5. Hamilton depression scale /17 Version (HAMD) score less than 10 points;
6. Memory decline at least 12 months, and the decline is progressive;
7. Brain MRI examination was done within 6 months before screening;
8. Neurological examination had no obvious signs (except due to AD disease or peripheral injury);
9. Females were postmenopausal (menopause beyond 24 weeks), or accepted the surgical sterilization, or women of childbearing age agreed to take effective contraceptive measures during the study. Women of childbearing age or menopausal time shorter than 24 weeks must do the urine pregnancy test and results to be negative during the screening period;
10. Subjects should have stable and reliable caregivers, or have frequent contact with caregivers (at least 4 days per week, at least 2 hours per day), caregivers will help patients to participate in the study. Caregivers must accompany the subjects in the study visit to provide valuable information for the NPI, ADCS-ADL and CIBIC-plus scales assessments;
11. Subjects have at least primary school education level, and have the ability to complete the determination of cognitive ability assessments and other tests;
12. The participants and legal guardian must sign informed consent.

Exclusion Criteria:

1. Brain MRI examination showed significant focal lesions, moderate-to-severe white matter lesions, and key parts lacunar infarction such as the thalamus, hippocampus, entorhinal cortex, cortical and subcortical gray matter nuclei;
2. Other type of dementia except AD;
3. Suffered from nervous system diseases (including stroke, optic myelopathy, Parkinson's disease, epilepsy, etc);
4. Psychotic patients, according to the DSM-5 criteria, include schizophrenia or other psychiatry disorders, bipolar disorder, major depression disorder, or delirium;
5. Abnormal laboratory test results: HBsAg and HBeAg and/or HbcAb positive and active stage of hepatitis B, liver function (ALT, AST) more than 1.2 times of the upper limit of the normal range, Cr exceeds the upper limit of normal, white blood cell count less than 4 x 109/L or platelet less than 100 x 109/L, hemoglobin less than 100g/L, blood glucose concentration of diabetic subjects (random) is more than 13.9mmol/L;
6. Systolic pressure was more than 160mmHg or less than 90mmHg, diastolic blood pressure was more than 100mmHg or less than 60mmHg;
7. With unstable or serious heart, lung, liver, kidney and hematopoietic system diseases (including unstable angina, myocardial infarction, uncontrolled asthma, gastric cancer, et al), or resting heart rate after 10 minutes of rest was less than 60 BPM, or QTc (QTc B (Bazett's correction value) or QTc F (Fridericia's correction value)) was equal or greater than 450msec, or with bundle branch block, the QTc B or QTc F was equal or greater than 480msec, or the researchers estimate there were abnormal EKG results which cannot be randomized to the study;
8. There was uncorrected of visual and auditory disturbances, and neuropsychological tests and scale assessments cannot be completed by the subject;
9. Subject was currently using Alzheimer's disease drugs and cannot be terminate the treatment;
10. Subjects that cannot take the test drug according to the prescription should be excluded;
11. Alcohol abuse or drug abuse;
12. Pregnant or lactating women;
13. Participated in other clinical pharmacological tests within 30 days before screening visit;
14. The researchers believe that the subject was impossible to complete the study;
15. Participants were employees of the study and immediate family members, employees of CRO company or sponsor and their immediate family members.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-09-16 (Estimated); Study Completion 2021-02-16 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive section (ADAS-Cog) | 26 weeks double-blind study and 28 weeks extention study
  The change of ADAS-Cog from baseline to endpoint among three arms.

SECONDARY OUTCOMES:
Clinician's Interview Based Impression of Change - plus (CIBIC+) | 26 weeks double-blind study and 28 weeks extention study
  The change of CIBIC+ from baseline to endpoint among three arms.
Activities of Daily Living (ADL) | 26 weeks double-blind study and 28 weeks extention study
  The change of ADL from baseline to endpoint among three arms.
Neuropsychiatric Inventory (NPI) | 26 weeks double-blind study and 28 weeks extention study
  The change of NPI from baseline to endpoint among three arms.

CONTACTS AND LOCATIONS:
Overall Officials: Shifu Xiao, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Other researchers should apply to the sponsor.